CLINICAL TRIAL: NCT05079126
Title: Double-Blind, Placebo-Controlled Study of Trans Sodium Crocetinate in Patients With Interstitial Lung Disease
Brief Title: Study of Trans Sodium Crocetinate in Patients With Interstitial Lung Disease
Acronym: ILD-DLCO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to, among other things, positive results from the 200-302 trial, the trial has been terminated early. Resources shifted to new 200-208 GBM trial using information gained from 200-302.
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100-601
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — trans-sodium crocetinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2.5 mg/kg Trans Sodium Crocetinate (Experimental): Subjects will receive a single IV bolus dose of 2.5 mg/kg TSC.
  Interventions: Drug: Trans Sodium Crocetinate
- Placebo (Placebo Comparator): Subjects will receive a single IV bolus dose of 7 mL Normal Saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trans Sodium Crocetinate — Single IV Bolus
  Arms: 2.5 mg/kg Trans Sodium Crocetinate
Drug: Placebo — Single IV Bolus
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled study of Trans Sodium Crocetinate (TSC) in patients with Interstitial Lung Disease (ILD), age 30-85 (inclusive). The primary objective of the study is to determine the effect of TSC on lung function as measured by diffusing capacity of the lungs for carbon monoxide (DLCO) in patients with ILD; the secondary objectives are to determine the effect of TSC on the 6-minute walk test (6MWT), heart rate recovery (HRR), and Borg Scale in patients with ILD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, age 30 to 85 years at screening
2. Able to provide informed consent and agree to adhere to all study visits and requirements
3. Females of childbearing potential must have a negative blood pregnancy test at screening and agree to use one of the accepted contraceptive regimens, or a double method of birth control during the study and at least 30 days after the last dose of study drug
4. Established diagnosis of ILD (clinical, radiographic, or histologic)
5. SpO2 ≥ 88% at rest by pulse oximetry while breathing ambient air
6. Free of any active cardiovascular or neuromuscular disease, at PI discretion
7. Clinically stable disease with no major medication changes in the last 4 weeks
8. Forced vital capacity (FVC) ≥ 45% of predicted (within past 6 months)
9. DLCO corrected for hemoglobin 30-90% of predicted, inclusive (within past 6 months)
10. Sars-CoV-2 negative at screening

Exclusion Criteria:

1. Known allergy to study medication
2. Pregnancy or lactation
3. Current smoker
4. Inability to perform pulmonary function testing
5. Active infection at screening or day of study visit
6. Known pulmonary hypertension (PH) requiring PH-specific treatment
7. AST/ALT ≥ 3x ULN and/or total bilirubin ≥ 2x ULN
8. Received any investigational medicine (IMP) within past 30 days
9. Surgery or hospitalization in past 3 months determined by the PI to be clinically relevant.
10. Current alcohol or substance abuse
11. Known active or latent hepatitis B or C
12. History of end-stage liver or renal disease
13. Positive COVID test anytime within 3 months of screening. Note:

    Patients who were previously vaccinated for COVID are allowed
14. History of venous thromboembolic disease
15. History of acute or chronic ophthalmologic conditions currently requiring treatment

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 30 minutes in DLCO after administration of a single dose of TSC versus placebo in patients with ILD | 30 minutes
  Compare the proportion of patients who achieve a prespecified level of improvement in DLCO 30 minutes after administration of the study drug (TSC or placebo) between the 2 randomized treatment arms.

SECONDARY OUTCOMES:
Change from baseline in 6MWT after administration of a single dose of TSC versus placebo in patients with ILD | 60 minutes
  Compare the proportion of patients who achieve a pre-specified level of improvement in 6 minute walk test (6MWT) after administration of the study drug (TSC or placebo) between the 2 randomized treatment arms.
Change from baseline in HRR after each 6MWT | 60 minutes
  Compare the proportion of patients who achieve a pre-specified level of improvement in heart rate recovery (HRR) after administration of the study drug (TSC or placebo) between the 2 randomized treatment arms.
Change from baseline in the Borg Scale after the 6MWT | 60 minutes
  Compare the proportion of patients who achieve a pre-specified level of improvement in the Borg dyspnea scale after administration of the study drug (TSC or placebo) between the 2 randomized treatment arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates, P.A., Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No